CLINICAL TRIAL: NCT00257608
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase IIIb Trial Comparing Bevacizumab Therapy With or Without Erlotinib After Completion of Chemotherapy With Bevacizumab for the First-Line Treatment of Locally Advanced, Recurrent, or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study Comparing Bevacizumab Therapy With or Without Erlotinib for First-Line Treatment of Non-Small Cell Lung Cancer (ATLAS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF3671g; BO20800 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Lung Cancer; ATLAS; Avastin; Tarceva
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: erlotinib HCl
- 2 (Placebo Comparator)
  Interventions: Drug: bevacizumab; Drug: placebo

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: placebo — Oral repeating dose
  Arms: 2
Drug: erlotinib HCl — Oral repeating dose
  Arms: 1

SUMMARY:
This is a Phase IIIb, multicenter, randomized, placebo-controlled trial to evaluate the safety and efficacy of chemotherapy+bevacizumab followed by bevacizumab+erlotinib versus bevacizumab+erlotinib placebo in subjects with locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically or cytologically confirmed NSCLC
* Advanced NSCLC or recurrent disease
* INR no greater than 1.3 and aPTT no greater than upper limits of normal (ULN) within 28 days prior to enrollment for subjects not on low molecular weight heparin or fondaparinux. Subjects on low molecular weight heparin or fondaparinux are not required to meet INR or aPTT limits. Chronic full-dose anticoagulation with warfarin is not permitted.
* 18 years of age or older
* For women of childbearing potential and sexually active men, use of an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to enrollment and for the duration of the study

Exclusion Criteria:

* Prior systemic chemotherapy in the metastatic setting
* Treatment with an investigational or marketed agent that acts by either EGFR inhibition or anti-angiogenesis mechanisms
* Pregnancy or lactation
* Any other medical condition, including mental illness or substance abuse, deemed by the clinician to be likely to interfere with a subject's ability to provide informed consent, cooperate, and participate in the study, or to interfere with the interpretation of the results
* Active infection or a fever within 3 days of enrollment
* Active malignancy other than lung cancer
* Radiation therapy to sites other than whole brain within 14 days prior to enrollment
* History of gross hemoptysis within 3 months prior to enrollment
* Known hypersensitivity to any of the components of cytotoxic chemotherapy combinations, bevacizumab, or tyrosine kinase inhibitors
* Inadequately controlled hypertension
* Unstable angina or New York Heart Association Grade II or greater CHF
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to enrollment
* History of myocardial infarction within 6 months prior to enrollment
* History of stroke within 6 months prior to enrollment
* Symptomatic peripheral vascular disease within 6 months prior to enrollment
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer, or bone fracture
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment; anticipation of need for major surgical procedure during the course of the study
* Current, recent, or planned participation in an experimental drug study other than this Genentech-sponsored bevacizumab/erlotinib study
* Progressive neurologic symptoms in subjects with a history of brain metastases
* History of significant vascular disease (e.g., aortic aneurysm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2006-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Strickland, M.D., Study Director — Genentech, Inc.
Locations (247):
- United States (177):
  - Sacred Heart Medical Onc Group, Mobile, Alabama
  - St. Edward Mercy Medical Ctr, Fort Smith, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Central Hem/Onc Medical Group, Alhambra, California
  - Comp Blood & Cancer Center, Bakersfield, California
  - South Bay Oncology, Campbell, California
  - Bay Area Cancer Research Grp, Concord, California
  - Pacific Onc & Hem Assoc, Encinitas, California
  - Pacific Coast Hem/Onc, Fountain Valley, California
  - Cancer Care Associates, Fresno, California
  - St. Jude Heritage Med Group, Fullerton, California
  - Ronald H. Yanagihara, Gilroy, California
  - Glendale Adventist Medical Ctr, Glendale, California
  - Scipps Clinic, La Jolla, California
  - Loma Linda Univ Medical Center, Loma Linda, California
  - Pacific Shores Medical Group, Long Beach, California
  - Kenmar Research Institute LLC, Los Angeles, California
  - UCLA Medical Ctr, Los Angeles, California
  - Sutter Gould Med Foundation, Modesto, California
  - North Valley Hem Onc Med Grp, Northridge, California
  - Hem Onc Med Grp Orange Cty, Orange, California
  - Medical Oncology Care Assoc, Orange, California
  - Ventura Co Hem-Onc Specialists, Oxnard, California
  - Wilshire Oncology Medical Grp, Pomona, California
  - Sutter Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Los Palos Oncology & Hem, Salinas, California
  - Kaiser Permanente, San Diego, California
  - Naval Medical Center, San Diego, California
  - Pacific Hematology Oncology, San Francisco, California
  - Kaiser Permanente Santa Teresa, San Jose, California
  - Sansum Medical Clinic, Inc., Santa Barbara, California
  - Santa Barbara Hem Onc Med Grp, Santa Barbara, California
  - Central Coast Medical Oncology, Santa Maria, California
  - The Angeles Clinic, Santa Monica, California
  - Redwood Regional Med Grp, Santa Rosa, California
  - Cancer Care Associates, Torrance, California
  - Mile High Oncology, Denver, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Washington Onc Hem Center PC, Washington D.C., District of Columbia
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Florida Wellcare Alliance, Inverness, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Mid-Florida Hem Oncology Ctr, Orange City, Florida
  - Integrated Comm Onc Network, Orange Park, Florida
  - Hematology Onc Treasure Coast, Port Saint Lucie, Florida
  - Phoebe Putney Cancer Center, Albany, Georgia
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Suburban Hem-Onc Associates, Lawrenceville, Georgia
  - Northwest Georgia Onc Centers, Marietta, Georgia
  - Chicagoland Hematology Onc, Arlington Heights, Illinois
  - Weiss-Strauss Oncology Center, Chicago, Illinois
  - LaGrange Oncology Associates, Geneva, Illinois
  - La Grange Oncology Associates, LaGrange, Illinois
  - Associates in Medical Oncology, Oak Lawn, Illinois
  - Onc Hem Assoc of Central IL, Peoria, Illinois
  - West Suburban Cancer Center, River Forest, Illinois
  - OSF St. Anthony Med Ctr, Rockford, Illinois
  - Community Hospital, Munster, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Hematology Oncology Associates, Bettendorf, Iowa
  - Siouxland Hem-Onc Assoc LLP, Sioux City, Iowa
  - Covenant Clinic, Waterloo, Iowa
  - Gajera & Patel, PLLC, Hopkinsville, Kentucky
  - Kentuckiana Cancer Center, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Consultants in Blood Disorders, Louisville, Kentucky
  - Owensboro Medical Health Sys, Owensboro, Kentucky
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - H&J Weinberg Cancer Institute, Baltimore, Maryland
  - Oncology Hematology Associates, Clinton, Maryland
  - Maryland Oncology/Hema PA, Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Caritas St. Elizabeth Med Ctr, Boston, Massachusetts
  - Lahey Clinic Med Ctr, Burlington, Massachusetts
  - Metrowest Cancer Center, Framingham, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Kalamazoo Hem & Onc, Kalamazoo, Michigan
  - Marquette General Health Sys, Marquette, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Virginia Piper Cancer Inst, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Freeman Cancer Institute, Joplin, Missouri
  - Missouri Cancer Center, PC, Saint Charles, Missouri
  - St. Louis Univ Care Center, St Louis, Missouri
  - Arch Medical Services, Washington, Missouri
  - Billings Clinic, Billings, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - NE Hematology Oncology, PC, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comp Cancer Centers of Nevada, Las Vegas, Nevada
  - Ctr for Cancer & Hem Disease, Cherry Hill, New Jersey
  - Forte, Attas & Schleider, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Central State Medical Center, Freehold, New Jersey
  - St. Barnabas Health Care Sys, Livingston, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Hematology Oncology Assoc SJ, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - San Juan Onco Assoc, Farmington, New Mexico
  - Zale P Bernstein MD - PP, Buffalo, New York
  - Bassett Cancer Center, Cooperstown, New York
  - Adriondack Cancer Care, Glen Falls, New York
  - BRANY, Great Neck, New York
  - Queens Cancer Center, Jamaica, New York
  - Crystal Run Health Care, Middletown, New York
  - NYU Medical Center, New York, New York
  - Mem Sloan Kettering Cancer Ctr, New York, New York
  - SUNY Upstate, Syracuse, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - NorthEast Medical Center, Concord, North Carolina
  - Moses Cone Reg Cncr Ctr, Greensboro, North Carolina
  - Emerywood Hematology Oncology, High Point, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Beaufort County Hospital, Washington, North Carolina
  - Summa Health System, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Onc/Hem Care Clin Trials LLC, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mid Ohio Onc Hematology Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Dayton Clinical Oncology Prog, Dayton, Ohio
  - Ohio Cancer Specialists, Mansfield, Ohio
  - Signal Point Hem/Oncology Inc, Middletown, Ohio
  - Toledo Community Hospital, Toledo, Ohio
  - Forum Health Cancer Care Ctr, Youngstown, Ohio
  - Providence Portland Med Center, Portland, Oregon
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Armstrong County Memorial Hosp, Kittanning, Pennsylvania
  - Hem Onc Assoc Phys Lancaster, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Assoc in Hematology Oncology, Upland, Pennsylvania
  - Lankenau Medical Office Bldg, Wynnewood, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Palmetto Hematology Oncology, Spartanburg, South Carolina
  - Erlanger Health Systems, Chattanooga, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - Jackson-Madsion County Hosp, Jackson, Tennessee
  - Clopton Clinic, Memphis, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt University Medical, Nashville, Tennessee
  - Lone Star Oncology Consultants, Austin, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Texas Cancer Associates, Dallas, Texas
  - Texas Hematology Oncology, Dallas, Texas
  - JPS Center for Cancer Care, Fort Worth, Texas
  - Univ of Texas Medical Branch, Galveston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - SW Vermont Healthcare Onc Asoc, Bennington, Vermont
  - Vermont Ctr Cancer Medicine, Colchester, Vermont
  - Community Cancer Center, Rutland, Vermont
  - Peninsula Cancer Institute, Newport News, Virginia
  - SW Virginia Hem Onc, Roanoke, Virginia
  - Cascade Cancer Center, Kirkland, Washington
  - Northwest Medical Specialists, Tacoma, Washington
  - Univ Physicians Internal Med, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Oncology Alliance, Glendale, Wisconsin
  - Dean Clinic, Madison, Wisconsin
  - Medical Consultants LTD, Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
- Argentina (9):
  - Hospital Pirovano, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Hospital Toru, Buenos Aires
  - CEMIC, Buenos Aires
  - Centro Oncologico de Cordoba, Córdoba
  - COIR, Mendoza
  - Instituto Medico Privado, Resistencia
  - Clinica Oncologica de Rosario, Rosario
  - ISIS Clinica Especializada, Sante Fe
- Australia (4):
  - Holy Spirit Hospital Northside, Chermside, QLD
  - Sunshine Coast Cancer Centre, Nambour, QLD
  - Sir Charles Gairdner Hospital, Nedlands, WA
  - Burnside War Memorial Hospital, Toorak Gardens, SA
- Belgium (2):
  - Cliniques Univ St Luc, Brussels
  - CHR Citadelle Liege, Liège
- Brazil (3):
  - Instituto de cancer Arnaldo, São Paulo, São Paulo
  - Instituto Nacional do Cancer, Rio de Janeiro
  - Hospital Das Clinicas, São Paulo
- Bulgaria (9):
  - Regional Oncodispensary, Plovdiv
  - Regional Oncodispensary, Rousse
  - Regional Oncodispensary, Shumen
  - Regional Oncodispensary, Sofia
  - UMHAT "Queen Joanna", Sofia
  - National Specialized Hospital, Sofia
  - Regional Oncodispensary, Stara Zagora
  - MHAT "St Marina", Varna
  - Regional Oncodispensary, Veliko Tarnovo
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (6):
  - Azienda Ospedaliera Univ, Genova
  - Ist Nazion per Ricerca Cancro, Genova
  - Univ degli Studi di Napoli, Napoli
  - Azienda Ospedaliera, Parma
  - Azienda Osper di Perugia, Perugia
  - Divisione Onc Med dell'Azienda, Udine
- Mexico (4):
  - Torre Medica Cristobal Colon, Acapulco
  - Inst Nacional de Cancerologia, Distrito Federal
  - ISSSTE Merida, Mérida
  - Hospital de Especialidades, Torreon, Coahuila
- Philippines (6):
  - Philippine General Hospital, Manila, Luzon
  - The Medical City, Pasig, Luzon
  - Veterans Memorial Medical Ctr, Quezon City, Luzon
  - Perpetual Succour Hospital, Cebu City, Visayas
  - Univ of Santo Tomas Hospital, Manila
  - St Luke's Medical Center, Quezon City
- Romania (3):
  - Centrul de Onc Medical Lasi, Iași
  - Spitalul Clinic Judetean Sibiu, Sibiu
  - Spitalul Judetean de Urgente, Suceava
- National Cancer Center, Singapore, Singapore
- Spain (7):
  - Corporacio Sanitaria Parc, Sabadell, Barcelona
  - Hospital de Cruces, Barakaldo
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario, San Cristóbal de La Laguna
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Clinico Universitario, Valencia
- Taiwan (3):
  - Taichung Veterans Gen Hosp, Dawan
  - China Medical Univ Hosp, Taichung
  - National Taiwan University, Taipei
- Thailand (5):
  - Bumrungrad International Hosp, Bangkok
  - National Cancer Institute, Bangkok
  - Pramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hosp, Chiang Mai
- Bristol Heamatology & Onc Ctr, Bristol, United Kingdom

REFERENCES:
- [Derived] Johnson BE, Kabbinavar F, Fehrenbacher L, Hainsworth J, Kasubhai S, Kressel B, Lin CY, Marsland T, Patel T, Polikoff J, Rubin M, White L, Yang JC, Bowden C, Miller V. ATLAS: randomized, double-blind, placebo-controlled, phase IIIB trial comparing bevacizumab therapy with or without erlotinib, after completion of chemotherapy, with bevacizumab for first-line treatment of advanced non-small-cell lung cancer. J Clin Oncol. 2013 Nov 1;31(31):3926-34. doi: 10.1200/JCO.2012.47.3983. Epub 2013 Oct 7. PMID 24101054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 14 countries between 10 January 2006 and 19 June 2009.
Groups:
- Bevacizumab + Chemotherapy: Participants received one of six chemotherapy regimens (Carboplatin + Paclitaxel or Carboplatin + Gemcitabine or Carboplatin + Docetaxel or Cisplatin + Gemcitabine or Cisplatin + Docetaxel / Cisplatin + vinorelbine) followed by Bevacizumab on Day 1 of each cycle up to 4 cycles.
- Bevacizumab + Placebo: Participants who completed four cycles of chemotherapy + bevacizumab received Bevacizumab 15 milligram per kilogram (mg/kg) intravenously (IV) on Day 1 of every 21-day cycle along with matched Placebo to Erlotinib orally daily.
- Bevacizumab + Erlotinib: Participants who completed four cycles of chemotherapy + bevacizumab received received IV dose of Bevacizumab 15 mg/kg on Day 1 of every 21-day cycle along with Erlotinib as 150 mg per day orally daily.
Period: Chemotherapy Phase
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Started | 1145 | 0 | 0
Completed | 769 | 0 | 0
Not Completed | 376 | 0 | 0
Not completed — Adverse Event | 138 | 0 | 0
Not completed — Disease progression | 139 | 0 | 0
Not completed — Unwillingness or inability to comply | 6 | 0 | 0
Not completed — Need for concomitant/ancillary therapy | 27 | 0 | 0
Not completed — Patient's decision to discontinue | 35 | 0 | 0
Not completed — Unrelated intercurrent illness | 3 | 0 | 0
Not completed — Physician Decision | 28 | 0 | 0
Period: Post Chemotherapy Phase
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Started | 0 | 373 | 370
Completed | 0 | 109 | 126
Not Completed | 0 | 264 | 244
Not completed — Adverse Event | 0 | 34 | 38
Not completed — Disease progression | 0 | 204 | 168
Not completed — Unwillingness or inability to comply | 0 | 4 | 5
Not completed — Need for concomitant/ancillary therapy | 0 | 5 | 5
Not completed — Patient's decision to discontinue | 0 | 4 | 8
Not completed — Unrelated intercurrent illness | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 8 | 11
Not completed — Sponsor's decision to terminate study | 0 | 1 | 0
Not completed — Not treated | 0 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab + Placebo: Participants received Bevacizumab 15 milligram per kilogram (mg/kg) intravenously (IV) on Day 1 of every 21-day cycle along with matched Placebo to Erlotinib orally daily
- Bevacizumab + Erlotinib: Participants received Bevacizumab 15 mg/kg IV on Day 1 of every 21-day cycle along with Erlotinib as 150 mg per day orally daily
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib | Total
Number analyzed (Participants) | 373 | 370 | 743
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (10.8) | 62.9 (10.3) | 62.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 177 | 354
  Male | 196 | 193 | 389

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the length of time from randomization until documented disease progression or death from any cause, whichever occurred earlier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Data presented until cut-off date 18 July 2008.
Time Frame: Approximately 3 years
Population: Intent to treat (ITT) population included all participants who were randomized during the post-chemotherapy phase.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Number analyzed (Participants) | 373 | 370
months | 3.7 [2.86 to 4.04] | 4.8 [4.14 to 5.52]
Statistical Analysis 1: Comparison: Bevacizumab + Placebo vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.0006, Log Rank; Hazard Ratio, log = 0.708, 95% CI 2-sided [0.580 to 0.864]

2. Secondary Outcome: Number of Participants With Prospectively Identified Treatment Emergent Adverse Events (TEAE) During Chemotherapy Phase
Description: Treatment-emergent adverse events were events between administration of study drug and up to 30 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.. Number of participants who had Grade >=3TEAEs of pulmonary hemorrhage, gastrointestinal (GI) perforation, arterial thromboembolic (ATE) events, proteinuria, congestive heart failure (CHF), and hypertension were presented. Data presented up to data cutoff 18 July 2008.
Time Frame: Approximately 3 years
Population: Safety-evaluable enrolled participants: All participants who enrolled and received at least one dose of chemotherapy or Bevacizumab. N= Number of participants analyzed.
Measure: Number; unit: participants
Groups:
- Carboplatin + Paclitaxel: Participants received Intravenous (IV) dose of Carboplatin at a dose based on an area under the concentration-time curve (AUC) of 6 milligram /milliliter (mg/mL) × minute (min) and Paclitaxel 200 milligram per square meter (mg/m^2) over 3 hours, respectively followed by Bevacizumab on Day 1 of each 21-day cycle up to 4 cycles.
- Carboplatin + Gemcitabine: Participants received IV dose of Carboplatin at a dose based on the AUC of 5 mg/mL × min on Day 1 of each 21-day cycle and Gemcitabine 1200 mg/m^2 on Day 1 and Day 8 followed by Bevacizumab of each 21-day cycle up to 4 cycles.
- Carboplatin + Docetaxel: Participants received IV dose of Carboplatin at a dose based on the AUC of of 6 mg/mL × min and Docetaxel 75 mg/m^2, respectively followed by Bevacizumab on Day 1 of each 21-day cycle up to 4 cycles.
- Cisplatin + Gemcitabine: Participants received IV dose of Cisplatin 80 mg/m^2 on Day 1 of each 21-day cycle and Gemcitabine 1000-1250 mg/m^2 on Day 1 and Day 8 followed by Bevacizumab of each 21-day cycle up to 4 cycles.
- Other: Included participants who received Cisplatin + Docetaxel or Cisplatin + vinorelbine, participants who received only one of the two chemotherapies planned followed by Bevacizumab of each 21-day cycle up to 4 cycles.
Arm/Group | Carboplatin + Paclitaxel | Carboplatin + Gemcitabine | Carboplatin + Docetaxel | Cisplatin + Gemcitabine | Other
Number analyzed (Participants) | 524 | 326 | 162 | 104 | 28
participants
  Pulmonary hemorrhage | 6 | 2 | 3 | 1 | 2
  GI perforation | 6 | 0 | 2 | 0 | 0
  ATE events | 8 | 6 | 2 | 1 | 0
  Proteinuria | 1 | 5 | 2 | 2 | 0
  CHF | 3 | 1 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Prospectively Identified Treatment Emergent Adverse Events (TEAE) During Post-Chemotherapy Phase
Description: Treatment-related adverse events are defined as new events that occur following subject entry into the study or events that worsen following study entry state and are judged by the investigator to be possibly, probably or definitely related to study medication. Pulmonary hemorrhage, GI perforation, ATE events, proteinuria, CHF, and hypertension were prospectively identified TEAEs of grade >=3. Data presented until cut-off date 28 January 2009.
Time Frame: Approximately 3 years
Population: Safety-evaluable randomized Participants: All randomized Participants who received at least one complete or partial dose of Bevacizumab + Erlotinib or Bevacizumab + Placebo. N= Number of participants analyzed.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Number analyzed (Participants) | 367 | 368
participants
  Pulmonary hemorrhage | 2 | 3
  GI perforation | 0 | 1
  ATE events | 5 | 8
  Proteinuria | 7 | 7
  CHF | 1 | 3
  Hypertension | 22 | 23

4. Secondary Outcome: Number of Participants With Any Adverse Events During Post-Chemotherapy Phase
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event. Data presented up to data cutoff 19 June 2009.
Time Frame: Approximately 3.5 years
Population: Safety-evaluable randomized Participants: All randomized Participants who received at least one complete or partial dose of Bevacizumab + Erlotinib or Bevacizumab + Placebo. N= Number of participants analyzed. At the time of the 28 January 2009 data cutoff, an additional 25 patients had been randomized.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Number analyzed (Participants) | 367 | 368
participants | 319 | 353

5. Secondary Outcome: Incidence of Study Treatment Discontinuation for Reasons Other Than Disease Progression in Chemotherapy Phase
Description: Participants who experienced disease progression were discontinued from the study. Data presented up to data cutoff (18 July 2008).
Time Frame: Approximately 3 years
Population: Enrolled participants: All participants who were enrolled in the study. N= Number of participants analyzed.
Measure: Number; unit: participants
Groups:
- Carboplatin + Paclitaxel: Participants received Intravenous (IV) dose of Carboplatin at a dose based on an area under the concentration time curve (AUC) of 6 milligram /milliliter (mg/mL) × minute (min) and Paclitaxel 200 milligram per square meter (mg/m^2) over 3 hours, respectively followed by Bevacizumab on Day 1 of each 21-day cycle up to 4 cycles.
Arm/Group | Carboplatin + Paclitaxel | Carboplatin + Gemcitabine | Carboplatin + Docetaxel | Cisplatin + Gemcitabine | Other
Number analyzed (Participants) | 524 | 326 | 162 | 104 | 29
participants
  Adverse Event | 54 | 40 | 22 | 14 | 8
  Concomitant/ancillary therapy | 13 | 6 | 5 | 1 | 2
  Patient's Decision to Discontinue | 16 | 6 | 8 | 5 | 0
  Investigator's Decision | 13 | 5 | 7 | 3 | 0
  Unwillingness or inability to comply with study | 4 | 0 | 0 | 1 | 1
  Unrelated intercurrent illness | 1 | 0 | 1 | 1 | 0

6. Secondary Outcome: Incidence of Study Treatment Discontinuation
Description: Participants in post-chemotherapy phase were discontinued from the study for the reasons other than disease progression. Data presented Up to data cutoff 18 July 2008.
Time Frame: Approximately 3 years
Population: Intent to treat (ITT) population included all participants who were randomized during the post-chemotherapy phase.. N= Number of participants analyzed.
Measure: Number; unit: participants
Groups:
- Bevacizumab + Placebo: Participants who completed four cycles of chemotherapy + bevacizumab received Bevacizumab 15 milligram per kilogram (mg/kg) intravenously (IV) on Day 1 of every 21-day cycle along with matched Placebo to Erlotinib.
  orally daily.
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Number analyzed (Participants) | 373 | 370
participants
  Bevacizumab: AE | 34 | 38
  Bevacizumab: Concomitant/ancillary therapy | 5 | 5
  Bevacizumab: Patient's Decision to Discontinue | 4 | 8
  Bevacizumab: Investigator's Decision | 8 | 11
  Bevacizumab: Unwillingness or inability to comply | 4 | 5
  Bevacizumab: Unrelated intercurrent illness | 0 | 1
  Bevacizumab: Sponsor's decision | 1 | 0
  Bevacizumab: Lost to follow-up | 0 | 1
  Erlotinib/placebo: AE | 22 | 48
  Erlotinib/placebo: Concomitant/ancillary therapy | 4 | 7
  Erlotinib/placebo:Patient's Decision | 5 | 10
  Erlotinib/placebo: Investigator's Decision | 6 | 12
  Erlotinib/placebo:Unwillingness/inability comply | 4 | 2
  Erlotinib/placebo: Unrelated intercurrent illness | 0 | 2
  Erlotinib/placebo: Sponsor's decision | 1 | 0
  Erlotinib/placebo: Lost to follow-up | 0 | 1

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the length of time from randomization to death.
Time Frame: Approximately 3.5 years
Population: Intent-to-treat population included all participants who were randomized during the post-chemotherapy phase.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Number analyzed (Participants) | 373 | 370
months | 13.3 [12.12 to 14.52] | 14.4 [12.29 to 18.60]
Statistical Analysis 1: Comparison: Bevacizumab + Placebo vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.5341, Log Rank; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.698 to 1.205]

ADVERSE EVENTS:
Time Frame: Up to 30 days after discontinuation of study treatment
Description: Safety-evaluable randomized participants who had received at least one complete or partial dose of bevacizumab or erlotinib/placebo.
Arm/Group | Bevacizumab + Placebo | Bevacizumab + Erlotinib
Serious Adverse Events (participants affected / at risk) | 63/367 | 86/368
Other Adverse Events (participants affected / at risk) | 288/367 | 341/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Placebo (N=367) | Bevacizumab + Erlotinib (N=368)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 0 | 5
Asthenia (General disorders) | 0 | 2
Death (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Hyperthermia (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Encephalitic infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Cranial neuropathy (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 5
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Placebo (N=367) | Bevacizumab + Erlotinib (N=368)
Anaemia (Blood and lymphatic system disorders) | 21 | 19
Abdominal pain (Gastrointestinal disorders) | 12 | 19
Constipation (Gastrointestinal disorders) | 33 | 34
Diarrhoea (Gastrointestinal disorders) | 72 | 188
Nausea (Gastrointestinal disorders) | 39 | 75
Stomatitis (Gastrointestinal disorders) | 9 | 27
Vomiting (Gastrointestinal disorders) | 26 | 38
Asthenia (General disorders) | 12 | 20
Chest pain (General disorders) | 24 | 18
Fatigue (General disorders) | 91 | 126
Mucosal inflammation (General disorders) | 3 | 26
Pyrexia (General disorders) | 9 | 20
Urinary tract infection (Infections and infestations) | 9 | 23
Weight decreased (Investigations) | 21 | 43
Anorexia (Metabolism and nutrition disorders) | 36 | 76
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 39
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 35 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 29
Dizziness (Nervous system disorders) | 18 | 23
Dysgeusia (Nervous system disorders) | 10 | 23
Headache (Nervous system disorders) | 45 | 38
Neuropathy peripheral (Nervous system disorders) | 25 | 28
Depression (Psychiatric disorders) | 10 | 32
Insomnia (Psychiatric disorders) | 13 | 23
Proteinuria (Renal and urinary disorders) | 21 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 63
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 42
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 | 40
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 26
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 | 58
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 44
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 21
Rash (Skin and subcutaneous tissue disorders) | 69 | 204
Hypertension (Vascular disorders) | 85 | 87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.